CLINICAL TRIAL: NCT05859529
Title: A Single-center, Randomized, Open-label, Parallel-controlled Study Was Conducted to Compare the Pharmacokinetics of JS002 When Delivered Subcutaneously Via a Prefilled Syringe Versus a Prefilled Autosyringe in Healthy Subjects
Brief Title: A Pharmacokinetic Study of JS002 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS002-008-BE
Record Dates: First submitted 2023-04-23; First posted 2023-05-16 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Health Volunteer

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental：JS002 AI (Experimental): The drug was administered by a single subcutaneous injection via AI
  Interventions: Drug: JS002
- Experimental：JS002 PFS (Active Comparator): The drug was administered by a single subcutaneous injection via PFS
  Interventions: Drug: JS002

INTERVENTIONS:
Drug: JS002 — The drug was administered by a single subcutaneous injection

SUMMARY:
This study was a single-center, randomized, open-label, single-dose, parallel-controlled trial design conducted in healthy adult subjects. Subjects were randomly assigned to 1 of 2 parallel treatment groups: treatment group A received a single subcutaneous injection of JS002 150 mg via PFS, and treatment group B received a single subcutaneous injection of JS002 150 mg via AI. Subjects were followed up to study day 85 for pharmacokinetic equivalence assessment of JS002. A total of 159 subjects were planned to be included in each group. After signing the informed consent form and completing the screening examination, subjects will be randomly assigned to treatment arm A or treatment arm B if eligible for inclusion.

The study period consisted of a screening period of up to 21 days and a follow-up period of 12 weeks (85 days). Subjects were admitted to the phase I clinical research unit the day before dose administration (day 1) and were not allowed to leave until all examinations and assessments were completed on day 6 after dose administration and were allowed to return to the clinical research center for follow-up visits on days 8,11,15,22,29,43,57,71, and 85.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers aged 18-45 years at screening;
2. have the ability to read and understand, voluntarily participate in the study, sign the written informed consent, and be able to complete the relevant procedures and examinations in accordance with the protocol;
3. the body mass index (BMI) at screening ranged from 19 to 26 kg/m2 (inclusive), with body weight ≥50kg for men and ≥45kg for women;
4. sitting blood pressure ≥ 90/60mmHg and < 140/90mmHg during screening;
5. serum LDL-C level ≥1.8mmol/L and < 4.9mmol/L at screening;
6. serum TG level < 2.8mmol/L at screening;
7. infertile, or fertile women willing to use strict and effective contraceptive methods throughout the study, in addition, fertile female subjects should have negative blood pregnancy test results during the screening period.

Exclusion Criteria:

1. Any history of use of Evolocumab and/or Alirocumab and other targeted drugs against PCSK9;
2. Use of any therapeutic or investigational biologics within 6 months before baseline (day 1);
3. Use of any medications or supplements that can alter blood lipids or affect lipid metabolism within 30 days before baseline (day 1), including but not limited to: Statins (such as atorvastatin, rosuvastatin, etc.), cholesterol absorption inhibitors (such as ezetimibe), probucol, cholic acid chelators (such as cholestyramine), traditional Chinese medicine (such as Xuezhikang), fibrates, high-purity fish oil preparations (or omega-3 fatty acids 1000 mg/ day), niacin preparations (niacin > 50 mg), etc.
4. Initiation of new vigorous exercise (e.g., long-distance running) or dietary control, or major modification of previous diet or lifestyle (e.g., exercise, smoking, and alcohol consumption) within 30 days before baseline (day 1). Creatine kinase (CK) ≥3 times the upper limit of normal value (ULN) on the day before randomization (day-1);
5. A history of allergy to biologics of mammalian origin (including monoclonal antibodies);
6. Subjects with allergic diseases or allergic constitution;
7. Patients with definite diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, endocrine system, and metabolic system that require medical intervention or other diseases that are not suitable for clinical trial (such as psychiatric history);
8. Donating ≥400 mL within 3 months before screening, or donating ≥200 mL within 1 month before screening, or receiving blood transfusion;
9. Participants who participated in other drug clinical trials within 3 months before screening;
10. Those who had taken any prescription drugs, over-the-counter drugs, herbal medicines, or health supplements within 2 weeks before screening;
11. Heavy smokers and drinkers (drinking 14 units of alcohol per week:1unit = beer 360 mL, or liquor 45 mL, or wine 150 mL; Smoking ≥5 cigarettes per day), or unable to abstain from smoking or drinking alcohol during the study period;
12. Had a history of drug abuse, or used drugs within 3 months before screening, or had a positive urine drug screening test during the screening period;
13. Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), treponema pallidum antibody and acquired immunodeficiency syndrome (HIV) antibody positive;
14. Abnormal chest X-ray (posterior-anterior view) and abdominal B-ultrasound results with clinical significance (non-clinically significant conditions such as irritability of gallbladder wall, hepatic cysts, intrahepatic calcifications, intrahepatic bile duct stones, slight fatty liver, etc., should be excluded).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
AUC0-last | 85 days
  Area under the time-concentration curve from time 0 to last time of quantifiable concentration
Cmax | 85 days
  Maximum Concentration

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 85 days
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in physical examination, vital signs, electrocardiogram, laboratory tests.
Tmax | 85 days
  Time to reach maximum concentration
t1/2 | 85 days
  Elimination half life
CL/F | 85 days
  Apparent clearance
Vz/F | 85 days
  Apparent volume of distribution
AUECday1-85 | 85 days
  Area under the effect curve (AUEC) for LDL-C through Day 1 to day 85
PCSK9 | 85 days
  Serum concentration of PCSK9
Immunogenicity | 85 days
  Incidence of antidrug antibodies (ADA)
Immunogenicity | 85 days
  Titer of ADA-positive samples, and incidence of neutralizing antibodies (Nab)

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China